CLINICAL TRIAL: NCT02362269
Title: Personalized Vitamin D Supplementation in European and African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-0047; A538500 (Other: UW Madison); SMPH\POP HEALTH SCI\POP HLTH (Other: UW Madison)
Record Dates: First submitted 2015-01-22; First posted 2015-02-12 (Estimated); Results first posted 2020-11-13 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): The control group will receive 2500 IU of vitamin D3 daily.
  Interventions: Dietary Supplement: Vitamin D
- Dosing Algorithm Group (Experimental): The dosing algorithm group will initially receive 1000, 2500, or 4000 IU of vitamin D3 daily based on the baseline 25(OH)D. This group's dosing may be adjusted at the 3-month visit.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Gelcaps containing 1000, 2500, and 4000 IU of vitamin D3 will be obtained from Tischon corporation (Westbury, NY). The gelcaps will be protected from light and not stored above 25° C. Participants will be instructed to take their vitamin D3 gelcaps with supper daily. Compliance with study supplementation will be documented by pill count at the time of each study visits.

SUMMARY:
The proposed study is a randomized, double-blind, controlled, multi-center clinical trial of six months of daily oral vitamin D3 (cholecalciferol). This study will randomize 334 community-dwelling post-menopausal women of European and African descent (~167 from each ancestry) in a 1:1 ratio between the control arm and the dosing algorithm arm using stratified block randomization with a block size of six and stratification by site (ancestry). The sample size of 334 includes 10% over-recruitment to allow for loss to follow-up. The European ancestry women will be seen in the Madison clinic and the African ancestry women will be seen in the Milwaukee clinic. The proposed study will focus on post-menopausal women because this is the subset of the population that both Dr. Engelman's and Dr. Binkley's preliminary data are drawn from. Moreover, 25(OH)D concentrations are typically lower in women and in older individuals, since production of vitamin D in the skin following sun exposure decreases with age. Therefore, this group of individuals is likely to benefit the most from vitamin D supplementation, especially when personalized based on biology using the proposed dosing algorithm.

DETAILED DESCRIPTION:
Potential volunteers will be screened by telephone. Those meeting all inclusion and no exclusion criteria will be invited to a screening study visit. At screening, informed consent will be obtained. The study team will then collect the following to determine study eligibility: basic demographic information (age, ancestry, and education); medical history; medication and supplement use; and blood for screening 25(OH)D and calcium tests. At baseline, participants will be randomly assigned to the control or dosing algorithm group. Both participants and study staff who have contact with the participants will be blinded to group assignment. Follow-up visits will occur at three and six months. At baseline and follow-up visits, height and weight will be measured and blood will be drawn for the vitamin D panel, calcium, and PTH. Blood for DNA and body composition will only be obtained at the baseline visit. Participants will be asked to return all unused study supplements and compliance will be assessed at each follow-up visit by pill count. The control group will receive 2500 IU of vitamin D3 daily while the dosing algorithm group will initially receive 1000, 2500, or 4000 IU daily, with the initial dosing based on the 25(OH)D at baseline, and the dosing may be adjusted at the 3-month visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, community-dwelling postmenopausal woman of self-reported European (Madison site) or African (Milwaukee site) descent
* Able and willing to sign informed consent
* Baseline serum 25(OH)D concentration of 10.0-29.9 ng/mL
* Willing to not alter the amount of their baseline vitamin D supplementation during the course of this study
* Willing to use sunscreen (SPF ≥15) when sun exposure of >15 minutes is expected during the months of May through September

Exclusion Criteria:

* Diagnosis of kidney or liver disease (organs that metabolize vitamin D)
* Current hypercalcemia (serum calcium ≥ 10.5 mg/dL) or other disorders that may affect vitamin D metabolism and predispose to hypercalcemia, i.e., sarcoidosis, active tuberculosis or other granulomatous disease.
* Other chronic diseases or conditions potentially affecting vitamin D metabolism or absorption (inflammatory bowel disease, cystic fibrosis, ulcerative colitis, and malabsorptive surgery)
* History of nephrolithiasis
* Current use of medications that affect vitamin D metabolism (glucocorticoids, anticonvulsants, antifungals, and HIV/AIDS medications)
* History of any form of cancer within the past two years with the exception of basal or squamous cell skin lesions, in situ tumors or thyroid cancer
* Terminal illness/on hospice
* Severe end-organ disease (e.g., cardiovascular, pulmonary, etc.), which may limit the ability to complete the study
* Treatment with high dose vitamin D (≥50,000 IU weekly) or any active metabolites of vitamin D, e.g., calcitriol, within six months of screening; current use of multiple vitamins and other vitamin D supplements will be allowed.
* Use of tanning beds or salons or unwillingness to utilize sunscreen during periods of sun exposure of 15 minutes or longer from May through September
* Planned trips/vacations likely to be associated with substantial amounts of sun exposure during the course of the study (i.e., more than 500 miles south of Madison/Milwaukee)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Engelman, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin Osteoporosis Clinical Research Program, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Dosing Algorithm Group
Started | 83 | 86
Completed | 82 | 80
Not Completed | 1 | 6
Not completed — Moved | 1 | 0
Not completed — Lost to Follow-up | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Dosing Algorithm Group | Total
Number analyzed (Participants) | 83 | 86 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.9) | 63.6 (6.7) | 63.5 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 86 | 169
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 82 | 86 | 168
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 15 | 29
  White | 69 | 71 | 140
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline 25(OH)Vitamin D [Mean (Standard Deviation); unit: ng/mL] | 26.4 (7.5) | 27.8 (7.6) | 27.0 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of the Dosing Algorithm in Achieving Total 25(OH)D as Measured by the Percentage of Participants Ending With Concentrations of 35-50 ng/mL
Description: To validate the proposed vitamin D3 dosing algorithm, a vitamin D panel consisting of serum concentrations of vitamin D3 (cholecalciferol; an indicator of vitamin D3 absorption), 25(OH)D3, 25(OH)D2, the C3-epimer of 25(OH)D3 and 24,25(OH)2D as well as an assay to directly measure free serum 25(OH)D will be run on all the blood samples collected at the baseline, 3 month and 6 month visits.
Time Frame: 3 and 6 months
Measure: Number; unit: percentage of participants in goal range
Arm/Group | Control Group | Dosing Algorithm Group
Number analyzed (Participants) | 82 | 80
percentage of participants in goal range
  3 Months | 61.3 | 58.5
  6 Months | 47.6 | 50.3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening through 6 Month study visit.
Arm/Group | Control Group | Dosing Algorithm Group
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/80
Serious Adverse Events (participants affected / at risk) | 2/82 | 3/80
Other Adverse Events (participants affected / at risk) | 0/82 | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=82) | Dosing Algorithm Group (N=80)
Hemorrhagic stroke (Cardiac disorders) | 1 (1) | 0 (0)
Hip replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Elective surgery
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Viral gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urothelial carcinoma (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT02362269/Prot_SAP_000.pdf